CLINICAL TRIAL: NCT04803721
Title: Interplay Between Immune and Metabolic Programs in Myelodysplastic Syndromes: Involvement in Leukemia Transformation and Therapeutic Targeting
Brief Title: Interplay Between Immune and Metabolic Programs in Myelodysplastic Syndromes
Acronym: IMET-MDS
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0481
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndromes; T-cells; metabolism
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient with a myelodysplastic syndrome: Patient over 18 years of age with a myelodysplastic syndrome (WHO 2016 classification) of low risk (LR= International Prognostic Scoring System (IPSS)-R<4.5) or high risk (HR=Revised International Prognostic Scoring System>4.5)
- Control patient: Healthy blood donor (regardless of age) Or Patient >60 years old, see at the geriatrics platform of the hospital la Grave (CHU of Toulouse), having expressed his non opposition to participate in the study

SUMMARY:
Myelodysplastic syndromes (MDS) are a pre-leukemic condition with an extremely poor prognosis despite current treatments that justify new therapeutic approaches. Various studies have described the potential involvement of both immune compartment and cellular metabolism in the pathophysiology of MDS. The aim of this study is to determine the specific immune and metabolic profiles of the different classes of MDS and to identify predictive markers of progression/survival/response to therapy.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are a pre-leukemic condition with an extremely poor prognosis despite current treatments. It is the most frequent haematological disorder after the age of 65. Different approaches targeting the immune compartment have been developed but preliminary results seem to show variable response rates to these therapeutic highlighting the heterogeneity of MDS and the need to identify detailed immune profiles that are predictive of disease progression and can help in treatment choices. It therefore seems essential to complement the knowledge of immune profiles with an understanding of the metabolic profiles of MDS patients, as well as the links between these profiles and changes associated with progression and/or treatment resistance, in order to consider new therapeutic pathways.

Fresh samples from patients with MDS will be used to perform flow cytometry mapping of immune populations, T-cell and blast cell metabolism. Subsequently, a study of energy metabolism will be conducted using an extracellular flow analyzer and a sensitivity test for certain molecules targeting metabolic pathways. If possible, samples will be taken at different times during the course of treatment, according to the therapeutic protocols: diagnosis, progression/transformation, during azacitidine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Patient over 18 years of age with a myelodysplastic syndrome (WHO 2016 classification) of low risk (LR=IPSS-R<4.5) or high risk (HR=IPSS-R>4.5);
  * Patient naïve to specific treatment of MDS;
  * Patient who expressed no opposition to participating in the study. ;
  * Patient affiliated with the social security system.
* Control:

  * over 18 years of age,
  * Sample from blood donation (regardless of age) Or Patient >60 years old, see at the geriatrics platform of the hospital la Grave (CHU of Toulouse),
  * having expressed his non opposition to participate in the study

Exclusion Criteria:

* Patients:

  * Myeloid disease other than MDS (including chronic myelomonocytic leukemia and MDS/SMP) ;
  * Ongoing treatments for MDS (excluding erythropoietin, granulocyte colony-stimulating factor and transfusions) ;
  * Medical conditions that may interfere with immune system testing: active cancer, active autoimmune disease, inflammatory conditions, immunosuppressive therapy. ; * Pregnant or breastfeeding women ; Patient's refusal ;
  * Person benefiting from a system of protection for adults (including guardianship, curators and safeguarding of justice)
* Control:

  * Medical conditions that may interfere with immune system testing: active cancer, active autoimmune disease, inflammatory conditions, immunosuppressive therapy. ; * Pregnant or breastfeeding women ;
  * Patient's refusal ;
  * Person benefiting from a system of protection for adults (including guardianship, curators and safeguarding of justice)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with a myelodysplastic syndrome (WHO 2016 classification) of low risk (LR=IPSS-R<4.5) or high risk (HR=IPSS-R>4.5)
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Immune and metabolic profiles will be evaluated by immunophenotyping | Day 0
  phenotypic study of one or more leukocyte sub-populations by flow cytometry

SECONDARY OUTCOMES:
Identification of time to progression/transformation and time to death | Day 0 and through study completion, an average of 1 year
  Clinical and biological data will be collected during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Comont, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- IUCT-Oncopole University Hospital, Toulouse, France